CLINICAL TRIAL: NCT06503302
Title: The Effect of Doppler Ultrasound on Calcified Tendinitis: a Double Blind, Randomized Controlled Trial
Brief Title: The Effect of Doppler Ultrasound on Calcified Tendinitis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Taipei Medical University Shuang Ho Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: TMU-IJRB-N202311060
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2024-07

CONDITIONS: Calcific Tendinitis of Shoulder
Keywords: Doppler ultrasound
MeSH Terms: conditions — Rotator Cuff Tear Arthropathy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Doppler ultrasound (Experimental): The physician will use Doppler function detection to check if calcifications are under active inflammation before ultrasound-guided injection.
  Interventions: Diagnostic Test: ultrasound Doppler function detection
- Without Doppler ultrasound (Active Comparator): The physician will only open the Doppler image in the non-calcified area for patient blinding before the ultrasound-guided injection.
  Interventions: Diagnostic Test: ultrasound Doppler function detection

INTERVENTIONS:
Diagnostic Test: ultrasound Doppler function detection — Doppler function detection is an ultrasound technique that measures and visualizes blood flow within an object, such as vessels and soft tissue. It can be used to check for the inflammation status of calcifications by detecting blood flow around the calcified areas before performing an ultrasound-guided injection.

SUMMARY:
Calcific tendinitis of the shoulder, is a self-limiting disease characterized by the deposition of calcium phosphate crystals in the rotator cuff tendons. Patients will develop complications such as decreased range of motion of the shoulder joint, and thus reducing their quality of life. The most common site of occurrence is 1.5-2 cm away from the supraspinatus tendon insertion site on the greater tuberosity. The primary treatment for calcific tendinitis is conservative, such as non-steroidal anti-inflammatory analgesics for pain relieving, extracorporeal shock wave therapy, subacromial steroid injections, ultrasound-guided barbotage technique for aspirating and washing out calcific deposits. Ultrasound is being used in calcified tendinitis for evaluating its size, location, quality, and also using the color Doppler ultrasonography to evaluate its reactive inflammatory changes. However, the use of color Doppler ultrasonography in diagnosing and treating a shoulder pain with calcification is not being concluded yet. Therefore, the aim of this study is to evaluate the efficacy of color Doppler ultrasonography in calcified tendinitis.

DETAILED DESCRIPTION:
Purpose: To evaluate the efficacy of color Doppler ultrasonography in calcified tendinitis.

ELIGIBILITY:
Inclusion Criteria:

1. chronic shoulder pain for more than 1 month
2. shoulder X-ray showed calcified deposit

Exclusion Criteria:

1. patient with needle phobia
2. patient with known allergy to medication like Triamcinolone and Lidocaine

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Need for a Second Ultrasound-Guided Injection | between three days to one week after the initial ultrasound-guided injection
  Whether a second ultrasound-guided injection is needed within a short period after the initial ultrasound-guided treatment, meaning whether significant improvement can be rapidly achieved after the first ultrasound-guided injection (defined as a reduction in pain index ≥50%).

SECONDARY OUTCOMES:
Pain Index (Visual Analogue Scale, VAS) | before treatment, between three days to one week after the initial ultrasound-guided injection, within the fourth week after the initial ultrasound-guided injection
  A simple and quick assessment method using a numerical scale from 0 to 10, where "0" represents no pain at all and "10" represents the most unbearable pain. The participant rates their own pain level.
Size of Calcification | before treatment, between three days to one week after the initial ultrasound-guided injection, within the fourth week after the initial ultrasound-guided injection
  Assessed using shoulder X-rays. The principal investigator will prescribe shoulder X-rays in the anteroposterior and lateral views during clinic visits. An outcome assessor will measure the calcification three times in each direction and calculate the average of the three measurements. The larger area from the two directions will be taken as the final measurement result.
Quick Disabilities of the Arm, Shoulder, and Hand (QuickDASH) Questionnaire | before treatment, between three days to one week after the initial ultrasound-guided injection, within the fourth week after the initial ultrasound-guided injection
  QuickDASH is a subset of 11 items from the 30-item DASH and is a self-reported questionnaire in which the response options are presented as 5-point Likert scales. At least 10 of the 11 items must be completed for a score to be calculated and the scores range from 0 (no disability) to 100 (most severe disability). This score was designed be useful in patients with any musculoskeletal disorder of the upper limb. It also consists of two optional modules: high-level sports/performing arts and work modules (4 items each, scored from 1 to 5).

CONTACTS AND LOCATIONS:
Overall Officials: Hung-Chou Chen, Principal Investigator — Taipei Medical University Shuang Ho Hospital
Locations (1):
- Taipei Medical University-Shuang Ho Hospital, Ministry of Health and Welfare, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Janeiro J, Barreira SC, Martins P, Ninitas P, Campos J, Fonseca JE. Ultrasound Features Associated With Shoulder Complaints: Calcifications Larger Than 6 mm in Young Patients and Positive Doppler Are Associated With Pain. Front Med (Lausanne). 2021 Nov 19;8:715423. doi: 10.3389/fmed.2021.715423. eCollection 2021. PMID 34869414
- [Background] Janeiro J, Barreira S, Martins P, Sarmento M, Campos J, Fonseca JE. Ultrasound findings and prognosis of shoulder pain: A role for Doppler signal? J Clin Ultrasound. 2023 Jun;51(5):837-844. doi: 10.1002/jcu.23436. Epub 2023 Jan 30. PMID 36715681
- [Background] Cesarec G, Martinec S, Cicak N. CALCIFIC TENDINOPATHY: CALCIUM DEPOSIT MORPHOLOGY DIRECTLY AFFECTS PAIN AND FUNCTION OF THE SHOULDER. Acta Clin Croat. 2020 Jun;59(2):270-276. doi: 10.20471/acc.2020.59.02.10. PMID 33456114
- [Background] Bazzocchi A, Pelotti P, Serraino S, Battaglia M, Bettelli G, Fusaro I, Guglielmi G, Rotini R, Albisinni U. Ultrasound imaging-guided percutaneous treatment of rotator cuff calcific tendinitis: success in short-term outcome. Br J Radiol. 2016;89(1057):20150407. doi: 10.1259/bjr.20150407. Epub 2015 Nov 26. PMID 26607641
- [Background] Patil P, Dasgupta B. Role of diagnostic ultrasound in the assessment of musculoskeletal diseases. Ther Adv Musculoskelet Dis. 2012 Oct;4(5):341-55. doi: 10.1177/1759720X12442112. PMID 23024711